CLINICAL TRIAL: NCT02055378
Title: the Effect of Low-Concentration Atropine Combined With Auricular Acupoint Stimulation in Myopia Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99-IRB-032-XD
Record Dates: First submitted 2014-02-02; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2012-12

CONDITIONS: Myopia
Keywords: myopia; atropine; anterior chamber depth; auricular acupoint; axial length
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- auricular acupoint stimulation (Experimental): Five auricular acupoints were selected for taping stimulation by using a 1-mm alloy ball by fingers three times a day, each time for five minutes over the five selected acupoints. Topical 0.125% atropine was given nightly.
  Interventions: Drug: Atropine; Device: auricular acupoint stimulation
- Atropine (Active Comparator): topical 0.125% atropine was given nightly during the study period.
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — topical 0.125% atropine eye drops
  Other Names: 0.125% atropine (Sinphar Pharmaceutical, Ilan, Taiwan)
Device: auricular acupoint stimulation — Five auricular acupoints (Shenmen, Xin, Yan, Mu 1 and Mu 2) Tapping stimulation was administered by using a 1-mm alloy ball (Magrain®; Sakamura, Kyoto, Japan) three times a day, each time for five minutes.
  Other Names: a 1-mm alloy ball (Magrain®; Sakamura, Kyoto, Japan)
  Arms: auricular acupoint stimulation

SUMMARY:
To compare the effect of myopia control between patients treated with low-concentration atropine eye drops combined with auricular acupoint stimulation and those treated with atropine alone.

DETAILED DESCRIPTION:
Myopia has been an increasing problem among school children, especially in Asian countries. High myopia is not only a refractive problem, but also a disease that can result in a number of sight-threatening complications such as macular degeneration, retinal detachment, glaucoma, and cataract. Atropine is a long-acting non-selective muscarinic antagonist that blocks accommodation by paralyzing ciliary muscles; it may affect remodeling of the sclera and suppress the elongation of axial length. Acupuncture and acupressure have been widely used in traditional Chinese medicine for thousands of years. Auricular acupoint stimulation by acupuncture or acupressure has been reported to improve visual acuity in myopic patients. Therefore, we want to compare the effect of myopia control between patients treated with low-concentration atropine eye drops combined with auricular acupoint stimulation and those who treated with atropine alone.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6 to 12 years with myopia, defined as spherical equivalent (SE) of -0.5 diopter (D) or less, were recruited from the outpatient clinics from January 2011 to June 2012.

Exclusion Criteria:

* (1) abnormal IOP (>21 mmHg) at presentation, (2) astigmatism or anisometropia of more than 1.5 D, (3) amblyopia or strabismus, (4) the presence of any related eyelid diseases, ocular diseases, or auricular diseases, (5) the presence of hemostatic disorders or other related major systemic diseases, (6) history of allergy to atropine, (7) previous or current use of contact lenses, bifocals, progressive lenses, or other forms of treatment for myopia.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the change in spherical equivalent (SE) | SE measured at 3, 6, 9, 12 months.
  We measured the myopic progression (change in SE) of all the participants for at least six months.

SECONDARY OUTCOMES:
axial length (AL) elongation, anterior chamber depth (ACD) and intraocular pressure(IOP) | AL, ACD, and IOP measure at 3, 6, 9, 12 months
  We measured the axial length (AL) elongation, anterior chamber depth (ACD) and intraocular pressure(IOP) of all the participants for at least six months.

CONTACTS AND LOCATIONS:
Overall Officials: Liao, MD, Study Chair — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taipei, New Taipei City, Taiwan